CLINICAL TRIAL: NCT02162901
Title: The Reach and Effectiveness of Technology-enhanced Diabetes Prevention Programs
Acronym: DiaBEAT-it
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Carilion Clinic (Other); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1R18DK091811-01A1 (NIH); 1R18DK091811-01A1 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Prevention
Keywords: Diabetes prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Choice-Class with IVR Calls (Experimental): Participants enrolled in this arm of the study will have chosen to attend one 2-hour class to be introduced to the educational intervention, and will then receive follow-up/support IVR calls for a period of 12 months.
  Interventions: Behavioral: Choice-Class with IVR Calls
- Choice-DVD with IVR calls (Experimental): Participants enrolled in this arm of the study will have chosen to watch a DVD at home to be introduced to the educational intervention, and will then receive follow-up/support IVR calls for a period of 12 months
  Interventions: Behavioral: Choice-DVD with IVR calls
- Random-Class with IVR calls (Experimental): Participants randomized to this arm of the study will be randomized a second time into one of three groups. Participants in this group will attend one 2-hour class to be introduced to the educational intervention, and will then receive follow-up/support IVR calls for a period of 12 months
  Interventions: Behavioral: Random-Class with IVR calls
- Random-DVD with IVR calls (Experimental): Participants randomized to this arm of the study will be randomized a second time into one of three groups. Participants in this group will be given a DVD to watch at home to be introduced to the educational intervention, and will then receive follow-up/support IVR calls for a period of 12 months
  Interventions: Behavioral: Random-DVD with IVR calls
- Random-Class only (Active Comparator): Participants randomized to this arm of the study will be randomized a second time into one of three groups. Participants in this group will attend one 2-hour class to be introduced to the intervention and will receive a workbook to use at home.
  Interventions: Behavioral: Random-Class only

INTERVENTIONS:
Behavioral: Choice-Class with IVR Calls — The intervention for this arm consists of an educational program which is an adaptation of the 16 lessons from the original Diabetes Prevention Program, both Core and After-Core sessions. After attending one 2-hour class to be introduced to the program and set goals, these lessons are delivered to the participant through 22 Interactive Voice Response telephone call over a period of 12 months.
  Arms: Choice-Class with IVR Calls
Behavioral: Random-Class with IVR calls — The intervention for this arm consists of an educational program which is an adaptation of the 16 lessons from the original Diabetes Prevention Program, both Core and After-Core sessions. After attending one 2-hour class to be introduced to the program and set goals, these lessons are delivered to the participant through 22 Interactive Voice Response telephone calls over a period of 12 months.
  Arms: Random-Class with IVR calls
Behavioral: Random-Class only — The intervention for this arm consists of an educational program which is an adaptation of the 16 lessons from the original Diabetes Prevention Program, both Core and After-Core sessions. After attending one 2-hour class to be introduced to the program and set goals, these lessons are delivered to the participant through a printed workbook.
  Arms: Random-Class only
Behavioral: Choice-DVD with IVR calls — The intervention for this arm consists of an educational program which is an adaptation of the 16 lessons from the original Diabetes Prevention Program, both Core and After-Core sessions. After watching a DVD at home to be introduced to the program and set goals, these lessons are delivered to the participant through 22 Interactive Voice Response telephone calls over a period of 12 months.
  Arms: Choice-DVD with IVR calls
Behavioral: Random-DVD with IVR calls — The intervention for this arm consists of an educational program which is an adaptation of the 16 lessons from the original Diabetes Prevention Program, both Core and After-Core sessions. After watching a DVD at home to be introduced to the program and set goals, these lessons are delivered to the participant through 22 Interactive Voice Response telephone calls over a period of 12 months.
  Arms: Random-DVD with IVR calls

SUMMARY:
The aim of this project is to evaluate the reach, effectiveness, and costs of two patient-centered, theory-based, technology-enhanced diabetes prevention programs to initiate and sustain weight loss among pre-diabetic adults (i.e. impaired fasting glucose or impaired glucose tolerance) within a health care setting. The overall aim is consistent with the NIDDK's Behavioral/Prevention Research Program's focus on individual, family, and community-based strategies for prevention of diabetes and its complications. While evidence of lifestyle interventions that increase physical activity and improve eating habits to achieve modest weight loss in delaying and preventing the onset of type 2 diabetes continues to mount, the translation of these interventions into effective programs to health care settings with modest resources remains a challenge. The proposed research project will conduct a pragmatic clinical trial that employs a hybrid Preference/Randomized Controlled Trial (RCT) designed to compare two technology-enhanced diabetes prevention programs in achieving objectively verified weight loss relative to a standard care control at comparatively lower costs. Adult patients (18 years of age and older) at risk for developing diabetes will be randomized to either the Choice group or the Randomization group. Those patients randomized to the Choice group (n=240) will have the opportunity to choose one of two programs to participate in: 1. A 2-hour Small-Group (SG) session, with automated interactive voice response (IVR) systems targeting personal action planning to support lifestyle change and weight loss over a period of 12 months; or 2. A DVD-based intervention with the same IVR follow-up. Those patients assigned to the RCT group (n=360) will be randomized to one of three groups: 1. SG/IVR; 2. DVD/IVR; or 3. Enhanced standard-care (SC). SC includes the referral to a currently offered pre-diabetes class. Primary outcome measures include weight loss, cost, and reach of each program. Secondary outcome measures include physical activity behavior; eating behavior; and process evaluation. It is hypothesized that both the SG/IVR and the DVD/IVR interventions will produce significantly greater amounts of weight loss at 6, 12, and 18 months following program initiation than SC but will not differ from one another. The investigators also hypothesize that the DVD/IVR will have broader reach and may be more cost-effective than SG/IVR or SC.

ELIGIBILITY:
Inclusion Criteria:

* age = or > 18 years
* BMI = or > 25

Exclusion Criteria:

* Patient's medical record contains ICD-9 codes for a diagnosis of any type of diabetes, congestive heart failure or coronary artery disease
* Pregnant or becomes pregnant during trial
* Contraindication to physical activity or weight loss
* No access to phone
* Does not speak or read English
* Patient has indicated "Do Not Contact" in Carilion patient record

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 months
  Weight as measured by clinical scale at baseline, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio A Almeida, PhD, MSW, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech Translational Obesity Research Center, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almeida FA, You W, Brito FA, Alves TF, Goessl C, Wall SS, Seidel RW, Davy BM, Greenawald MH, Hill JL, Estabrooks PA. A randomized controlled trial to test the effectiveness of two technology-enhanced diabetes prevention programs in primary care: The DiaBEAT-it study. Front Public Health. 2023 Feb 24;11:1000162. doi: 10.3389/fpubh.2023.1000162. eCollection 2023. PMID 36908422